## APPENDIX D Study Protocol Class Procedures

## Yoga for a Healthy Heart Protocol

| Week 8 | Week 7 | Week 6 | Weck 5 | Week 4 | Week 3 | Week 2 | Week 1 | |
|---|---|---|---|---|---|---|---|---|
| Mini and Medi-<br>Cog, Perceived<br>Stress Scale, BP | Pre-Class BP | Pre-Class BP | Pre-Class BP | Pre-Class BP | Pre-Class BP | Pre-Class BP | Mini and Medi-<br>Cog, Perceived<br>Stress Scale, BP | Assessment |
| Chair-based yoga | Chair-based yoga | Chair-based yoga | Chair-based yoga | Chair-based yoga | Chair-based yoga | Chair-based yoga | Chair-based yoga | Yoga physical practice |
| Full diaphragmatic breathing with one to two ratio; ujjayii | Full diaphragmatic breathing with one to one ration | Segmental diaphragmatic breathing stage two | Segmental diaphragmatic breathing stage one; add clavicular | Natural breath awareness; thoracic, abdominal breathing | Natural breath awareness; thoracic, abdominal breathing | Natural breath awareness; abdominal breathing | Natural breath<br>awareness;<br>abdominal<br>breathing | Yoga Breathing<br>Practice |
| Yoga Nidra and Ajapa visualization with mantra "I am" with positive | Yoga Nidra and Ajapa visualization with mantra "I am" | Yoga Nidra | Yoga Nidra | Yoga Nidra | Yoga Nidra | Yoga Nidra | Yoga Nidra | Yoga Meditation |
| Home Program;<br>Self-discípline;<br>Conclusion of<br>class | Energy conservation; acceptance | Energy<br>conservation; self-<br>study | Awareness of<br>breath with<br>movement; Non-<br>excess concept | Awareness of perceived effort; non attachment | Awareness of digestion and posture; simplicity | Awareness of breathing pattern and posture; truthfulness | Joint protection; "Do no harm" | Discussion with class theme |
| Post-class BP | Post-class BP | Post-class BP | Post-class BP | Post-class BP | Post-class BP | Post-class BP | Post-class BP | Assessment |